CLINICAL TRIAL: NCT01278277
Title: A Novel Therapeutic Strategy Targeting Photoreceptor Oxidative Damage in ABCR-related Retinal Degenerations
Brief Title: Saffron Supplementation in Stargardt's Disease
Acronym: STARSAF02
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Benedetto Falsini, Associate Professor Ophthalmology, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STARSAF02
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Retinal Degeneration; Genetic Disease; Single-Gene Defects; Macular Dystrophy
Keywords: Stargardt disease; macula; electroretinogram; saffron
MeSH Terms: conditions — Retinal Degeneration; Genetic Diseases, Inborn; Macular Degeneration; Stargardt Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo supplementation (Placebo Comparator): patients will be assigned, in a cross-over design, to placebo or supplement administration
  Interventions: Other: placebo
- Saffron (Active Comparator): Saffron Supplementation 20 mg/die
  Interventions: Dietary Supplement: Saffron supplementation

INTERVENTIONS:
Dietary Supplement: Saffron supplementation — Saffron supplementation 20 mg
  Other Names: Zaffit Special
  Arms: Saffron
Other: placebo — placebo supplementation
  Arms: placebo supplementation

SUMMARY:
The general area of research in which this project has been designed is that of retinal degeneration related to mutations in the ABCR gene, responsible of Stargardt disease/fundus flavimaculatus retinal dystrophy (STD/FF). STG/FF is one of the major causes of vision impairment in the young age. STG/FF originates typically from the dysfunction and loss of cone and rod photoreceptors, developing through a photo-oxidative mechanism. The major disease locus is the central retina, i.e. the macula, whose neurons have the highest density and underlie critical functions such as visual acuity, color vision and contrast sensitivity. There is currently no cure for STG/FF. Recent experimental findings indicate that Saffron, derived from the pistils of Crocus Sativus, may have a role as a retinal neuro-protectant against oxidative damage. The stigmata of Crocus sativus contain biologically high concentrations of chemical compounds including crocin, crocetin, whose multiple C=C bonds provide the antioxidant potential. In addition it is well known that this compound is safe and free of adverse side effects. The aim of this research is to investigate the influence of short-term Saffron supplementation on retinal function in STG/FF patients carrying ABCR mutations. The macular cone-mediated electroretinogram (ERG) in response to high-frequency flicker (focal flicker ERG) will be employed as the main outcome variable. Secondary outcome variable will be the psychophysical cone system recovery after bleaching.

DETAILED DESCRIPTION:
Research Plan Background Stargardt disease (STGD/FFM) is the most common hereditary recessive macular dystrophy (Blacharski, 1988) characterized by juvenile to young adult onset, central visual impairment, progressive bilateral atrophy of the macula and retinal pigment epithelium (RPE), with a frequent appearance of orange/yellow flecks distributed around the macula and/or the mid retinal periphery (Noble and Carr, 1971). A clinically similar retinal disorder, fundus flavimaculatus (FFM), often displays later ages of onset and slower progression. It has been suggested and demonstrated (Allikmets et al., 1997) that STGD and FFM represent allelic disorders. Mutations in the gene encoding an ATP-binding cassette (ABC) transporter (ABCR), mapping to chromosome 1p13-p21, have been found to be responsible of STGD (Allikmets et al., 1997). The ABCR gene is expressed exclusively and at high levels in the retina, in both rod and cone photoreceptors (Molday et al., 2000). A recent study by Weng et al. (1999) , investigating the molecular mechanisms underlying photoreceptor degeneration in ABCR knock-out mice, proposed that photoreceptors die as a consequence of 'poisoning' of the RPE by lipofuscin accumulation and loss of the RPE support role. Accumulation within the RPE cells of a compound, A2E, forming from condensation of phosphatydilethanlolamine and the all-trans-retinal released from photoactivated rhodopsin (Sparrow et al., 2000), probably leads in vivo to an increased absorption of blue lights and to phototoxic RPE cell damage. The mutation-induced disease may affect both rod and cone photoreceptors, at relatively early stages. In vitro studies (Sun and Nathans, 2001) also demonstrated that the ABCR itself is an efficient target of all-trans-retinal-mediated photooxidative damage.

Clinically, many reports have documented an abnormal functioning of both macular and peripheral cones, as well as rods, in STGD/FFM (Moloney et al., 1983; Lachapelle et al., 1990). There is also evidence (Lois et al., 2001) that STGD/FFM may be associated with different patterns of retinal dysfunction, with a selective involvement of macular function, or more widespread dysfunction involving cone and/or rod function, showing intrafamilial consistency. Characteristic abnormalities of dark adaptation (Aleman et al., 1999), involving a delayed post-bleach recovery, to the baseline sensitivity, of the last branch of the adaptation curve have been also described. Similar abnormalities in rod dark adaptation have been recently found in a mice heterozygous for a null mutation in the ABCR gene (Mata et al., 2001). Clinical evidence (Parisi et al., 2002) indicates that also the recovery of cone sensitivity after bleaching is severely impaired in STG/FF, suggesting that profoundly altered retinoid recycling, leading to photoxidative damage, specifically occurs in cone photoreceptors.

Recent experimental findings (Maccarone et al., 2008) indicate that Saffron, derived from the pistils of Crocus Sativus, may have a role as a retinal neuro-protectant against oxidative damage. Indeed, Saffron has been shown to be protective, for both morphology and function, in a rat model of light-induced photoreceptor degeneration. In this model, cell death is thought to result from oxidative stress induced by prolonged increase in oxygen tension and photooxidation. Saffron is an attractive candidate to be tested because the stigmata of Crocus sativus contain biologically high concentrations of interesting chemical compounds including crocin, crocetin (Giaccio, 2004), whose multiple C=C bonds give the antioxidant potential. Not to mention that its centuries-long use as spice, with no known ill effects increases the confidence in secure applicability. In addition it has been recently reported (Ochiai et al., 2007) that crocins are able to activate metabolic pathways to protect cells from apoptosis and to reduce light induced death in isolated photoreceptors (Laabich et al., 2006) , while crocetin (Giaccio, 2004) increases oxygen diffusivity through liquids, such as plasma. Considering the high metabolic rate of photoreceptors, the availability of oxygen may be a critical factor in protecting them from death. In addition, Kanakis et al. (Kanakis et al, 2007) showed that metabolites of antioxidant flavonoids bind directly to DNA and induce its partial conformation to beta-DNA, thereby protecting the cell from damage. Based on these observation it comes clear that Saffron extract does not act as a simple antioxidant. The peculiar characteristics of Saffron components support the hypothesis of an involvement of very different ways of action going from antioxidant activity to direct control of gene expression. These components may act in humans as protective agents against oxidative damage for the ageing retina, and may repair early photoreceptor damage associated with STG/FF, whose disease patho-physiology has been linked by experimental studies (Mata et al, 2001) to light-induced oxidative damage to the outer retina. In STG/FF eyes, at early disease stages, the normal number of cone photoreceptors is partially retained, although the cells might be dysfunctional. As a result of the rescuing effects of Saffron, the pool of damaged but viable photoreceptors could increase its response, resulting in improved retinal sensitivity.

The objective of the present project is to evaluate whether Saffron supplementation has a beneficial neuro-protective effect for the damaged retinas as consequence of ABCR mutation-STD/FF.

Clinical Protocol Patients A group of 30 STG/FF patients (14 males, 16 females, age range: 15-68 years) will be included in this study. Patients will meet the following inclusion criteria: 1. Macular and peripheral retinal degeneration with typical funduscopic lesions (retinal flecks) and a cone-rod pattern of retinal dysfunction, as determined by standard Ganzfeld electroretinography and dark-adapted fundus perimetry, and classic fundus appearance, 2. Relatively preserved central retinal function (visual field by Goldmann V/4e > 30°, corrected EDTRS visual acuity > 20/80) and stable central fixation as determined by a Visuskope, 3. Known genotype or genotype under study, 4. At least four follow-up clinical examination over the past three years, 5. No or minimal ocular media opacities, 6. No concomitant ocular (e.g. glaucoma, amblyopia) or systemic diseases. Informed consent for all patients and controls will be obtained after the aims and procedures of the study will be explained in detail.

Treatment and Testing Schedule The patients will be divided into two groups: 15 will treated with oral supplementation of a daily dose of Saffron for 90 days, and 15 will undergo placebo treatment during the same period. At the end of a 90 days period the patients will be crossed-over and assigned respectively to placebo or Saffron supplementation. In all patients, clinical examination, including visual acuity testing with a calibrated standard Snellen chart and fundus examination by direct and indirect ophthalmoscopy, and FERG testing will be performed at the study entry (baseline) and after 180 days of treatment or placebo. In all cases, compliance will be judged by telephone interview and pill counts. Adverse side effects will be reported.

Electrophysiological Methods FERG testing will be performed according to a previously published technique (Falsini et al., 2000). Briefly, ERGs will be elicited by the LED-generated sinusoidal luminance modulation of a circular uniform field (18° in diameter, 80 cd/m2 mean luminance, dominant wavelength: 630 nm), presented at the frequency of 41 Hz on the rear of a ganzfeld bowl, illuminated at the same mean luminance as the stimulus. A series of FERG responses will be collected at different modulation depths [quantified by the Michelson luminance contrast formula: 100%*(Lmax -Lmin)/(Lmax +Lmin), where Lmax and Lmin are maximum and minimum luminance, respectively] between 16.5% and 93.8% in 0.1 to 0.3 log unit steps. FERG signals will be acquired in sequence for six values of modulation depth between 16.5 to 93.5%, presented in an increasing order. For each patient FERG log amplitudes will be plotted as a function of log modulation depth. The resulting function's slope will be determined by a linear regression. From the same regression line, FERG threshold will be estimated from the value of log modulation depth yielding a criterion amplitude, corresponding to a S/N ratio of 3.

Psychophysics An increment threshold technique will be used to evaluate the recovery of cone system sensitivity after bleaching exposure. Psychophysical threshold will be determined at the paracentral visual field locations with preserved visual sensitivity, by presenting a 0.5 sec flashing light on a light adapting background of 20 cd/sqm. Following baseline assessment, the threshold intensity for the flashed light will be measured and plotted as a function of time, following 30 sec exposure to an adapting light (delivered in Maxwellian view by means of a calibrated indirect ophthalmoscope) whose intensity is estimated bleach approx 30% of the cone photopigment. The resulting dynamic recovery function, fitted by an exponential function, describes the sensitivity recovery of the photopic system following bleaching, and reflects either the rate of free opsin inactivation or photopigment synthesis. A computer-controlled system, employing a commercially available apparatus, has been developed (Fadda et al., 2001) for measuring bleaching adaptation of the cone system.

Statistical Analysis Sample size estimates of patients for this study will be based on previous investigations (Parisi et al., 2001) where the between- and within-subjects variability (expressed as data SD) of FERG parameters was determined in STG/FF patients. Assuming between- and within-subjects SDs in FERG amplitude and phase of 0.1 logmicroV and 20 degrees, respectively, the sample sizes of patients assigned to both Saffron and placebo provide a power of 80%, at an alpha = 0.05, for detecting in each group a test-retest difference (i.e. 90 days minus baseline test) of 0.1 logmicroV (SD: 0.1) and 30 degrees (SD: 20) in amplitude and phase, respectively. Results will be analyzed by multivariate statistics (multivariate analysis of variance for repeated measures, MANOVA). In all the analyses a p < 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Macular and peripheral retinal degeneration with typical funduscopic lesions (retinal flecks)
* Relatively preserved central retinal function
* Known genotype or genotype under study

Exclusion Criteria:

* absence of a rod-cone pattern of dysfunction
* acuity less than 0.1
* Unknown genotype

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Focal electroretinogram (FERG) | six months
  ERGs will be elicited by the LED-generated sinusoidal luminance modulation of a circular uniform field (18° in diameter, 80 cd/m2 mean luminance, dominant wavelength: 630 nm), presented at the frequency of 41 Hz on the rear of a ganzfeld bowl, illuminated at the same mean luminance as the stimulus.

SECONDARY OUTCOMES:
Psychophysical recovery of cone system sensitivity after bleaching | six months
  Psychophysical threshold will be determined at the paracentral visual field locations with preserved visual sensitivity, by presenting a 0.5 sec flashing light on a light adapting background of 20 cd/sqm. Following baseline assessment, the threshold intensity for the flashed light will be measured and plotted as a function of time, following 30 sec exposure to an adapting light (delivered in Maxwellian view by means of a calibrated indirect ophthalmoscope) whose intensity is estimated bleach approx 30% of the cone photopigment.

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Falsini, MD, Principal Investigator — Catholic University of the Sacred Heart; Marco Piccardi, MD, Principal Investigator — Catholic University of the Sacred Heart; Silvia Bisti, PhD, Study Director — University of L'Aquila
Locations (1):
- Policlinico A. Gemelli, Rome, Italy

REFERENCES:
- [Background] Falsini B, Piccardi M, Minnella A, Savastano C, Capoluongo E, Fadda A, Balestrazzi E, Maccarone R, Bisti S. Influence of saffron supplementation on retinal flicker sensitivity in early age-related macular degeneration. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6118-24. doi: 10.1167/iovs.09-4995. Epub 2010 Aug 4. PMID 20688744
- [Derived] Piccardi M, Fadda A, Martelli F, Marangoni D, Magli A, Minnella AM, Bertelli M, Di Marco S, Bisti S, Falsini B. Antioxidant Saffron and Central Retinal Function in ABCA4-Related Stargardt Macular Dystrophy. Nutrients. 2019 Oct 15;11(10):2461. doi: 10.3390/nu11102461. PMID 31618812